CLINICAL TRIAL: NCT00284479
Title: The Effect of a Worksite Based Walking Programme on Cardiovascular Risk in Previously Sedentary Civil Servants
Brief Title: The Effect of Walking on Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Murtagh/Murphy 2004
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2003-01

CONDITIONS: Sedentariness
Keywords: walking intervention; cardiovascular risk; inflammatory markers; aerobic fitness; fatness

INTERVENTIONS:
Behavioral: Walking 45 mins 2x p.w.

SUMMARY:
The purpose of this study was to investigate the effects of an 8 week program of walking for 45 minutes, twice a week, on fitness, body composition , blood pressure and blood markers of cardiovascular risk. We hypothesised that this 90 minutes of walking per week would result in measurable increases in fitness and reductions in body fat, resting blood pressure and improved blood lipid profiles.

DETAILED DESCRIPTION:
Current physical activity guidelines suggest that every adult should accumulate 30 minutes or more of moderate intensity physical activity on most days of the week. However, compliance with these guidelines requires considerable commitment in terms of time spent exercising per week (> 150 minutes) and this may deter individuals from starting an exercise programme. Accordingly, randomised controlled trials are needed to evaluate the effects of smaller volumes of exercise on health.

37 civil servants (24 women) aged 41.5 + 9.3 years, were randomly assigned to either two 45 minute walks per week (walking group) or no training (control group). Aerobic fitness, body composition, blood pressure (BP), CRP and lipoprotein variables were measured at baseline and following 8 weeks. Steps counts were measured at baseline and during weeks 4 and 8 of the intervention

ELIGIBILITY:
Inclusion Criteria:

Member of staff at the Northern Ireland Civil Service

Exclusion Criteria:

Physically active (defined as compliance with current physical activity guidelines (Pate, 1995), age > 65 years, resting BP > 159/99 mm Hg, total cholesterol > 6.2 mmol•L-1, fasting blood glucose > 7.0 mmol•L-1, body mass index (BMI) > 34.9 kg•m-2, current cigarette smokers, individuals with cardiovascular, pulmonary or metabolic disease, pain or discomfort in the chest, dizziness or heart murmur.

individuals taking medication known to interfere with lipid metabolism, females who were pregnant or planning to become pregnant in the following five months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-05; Study Completion 2003-01

PRIMARY OUTCOMES:
Aerobic Fitness
Resting Blood Pressure
Body Fatness
Blood Lipids
C-reactive Protein

CONTACTS AND LOCATIONS:
Overall Officials: Marie H Murphy, Study Director — University of Ulster at Jordanstown
Locations (1):
- University of Ulster, Newtownabbey, Co Antrim, United Kingdom

REFERENCES:
- [Result] Murphy MH, Murtagh EM, Boreham CA, Hare LG, Nevill AM. The effect of a worksite based walking programme on cardiovascular risk in previously sedentary civil servants [NCT00284479]. BMC Public Health. 2006 May 22;6:136. doi: 10.1186/1471-2458-6-136. PMID 16716211